CLINICAL TRIAL: NCT03664427
Title: Pharmacogenetics of Veno-Occlusive Disease (VOD) in Children With Haematological Stem Cell Transplantation (HSCT)
Brief Title: Pharmacogenetics of VOD in Children With HSCT
Acronym: MVO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI16025J
Record Dates: First submitted 2018-07-09; First posted 2018-09-10 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2021-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients with VOD: paediatric patients with Veno-Occlusive Disease (VOD) complicating haematological stem cell transplantation
- Group 2: matched controls: Paediatric patients defined as matched controls without veno-occlusive disease complicating haematological stem cell transplantation

SUMMARY:
This project aims to identify common pharmacogenetic biomarkers predisposing children with cancer to develop hepatic VOD during their cancer treatment including HSCT. The impact of VOD occurrence and significant biomarkers will also be evaluated on outcome at day 100 and one year after HSCT. It should help to highlight factors that can contribute to the initiation of hepatic VOD.

Understanding mechanisms of this toxicity and to know individual parameters of disease susceptibility becomes an important issue in the care of these children. The ultimate goal of research in this area would be to develop a personalized predictive medicine and, hopefully, prevent the occurrence of VOD from a therapeutic adaptation to each patient according to his pharmacogenetic profile (adapted prophylaxis, dose adjustment, drug combinations ...). A prospective identification of patients at risk of hepatic VOD will increase the safe use of anticancer.

DETAILED DESCRIPTION:
Hematopoietic stem cells transplantation (HSCT) in children with cancer is source of veno-occlusive disease (VOD). This complication is unpredictable and serious by involving the vital prognosis of the child. In addition, this complication may affect the patient's quality of life and have serious long-term sequelae. The incidence varies from 15 to 60% and the mortality is greater than 60% after severe VOD. The risk factors of occurrence of these complications are, to date, unknown except for a susceptibility to some therapeutic (busulfan, radiotherapy ...). Pharmacogenetic aspects of hepatic VOD susceptibility are supposed and targeted screening supported this hypothesis. But pharmacogenetic predisposition to VOD was never explored with as many polymorphisms and considering the whole exome.

ELIGIBILITY:
Inclusion Criteria:

* Children with cancer aged less than 18 years old treated for their first HSCT between 2000 and 2011 in France.
* Patients are selected from the database ProMise regarding pediatric patients treated in any center of the French Society of Stem Cell transplantation (SFGM).
* Clinical data (age, sex, initial pathology, conditioning treatment, type of graft cells, VOD occurence or not, survival status at 100 days and 1 year after transplantation) were extracted from this database.

Exclusion Criteria:

-

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study concerns children with cancer aged less than 18 years treated for their first HSCT between 2000 and 2011 in France.
Sampling Method: Probability Sample
Enrollment: 436 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Pharmacogenetic biomarkers | 12 months
  The pharmacogenetic analysis will be conducted by a whole exome genotyping approach with Microarrays Illumina "Human Omni2.5-8 v1.3" (exploring more than 2,600,000 genetic variants covering the entire genome with more than 300,000 genetic biomarkers within exons).

SECONDARY OUTCOMES:
Survival status at 100 days post HSCT | 100 days
  Survival at 100 days post-HSCT will be evaluated according to the occurrence or not of VOD
Survival status at 1 year post HSCT | 12 months
  Survival at 1 year post-HSCT will be evaluated according to the occurrence or not of VOD

CONTACTS AND LOCATIONS:
Overall Officials: Evelyne Jacqz-Aigrain, MD, PhD, Principal Investigator — APHP
Locations (1):
- Robert Debre Hospital, Paris, France